CLINICAL TRIAL: NCT02842814
Title: Evaluation and Prediction of Relapse Risk After Glucocorticoid Withdrawal in Patients With Stable Systemic Lupus Erythematosus: An Open-labeled Multi-centric Randomized Controlled Study From China
Brief Title: Prediction of Relapse Risk in Stable Systemic Lupus Erythematosus
Acronym: PRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Xiangya Hospital of Central South University (Other); Shengjing Hospital (Other); People's Hospital of Xinjiang Uygur Autonomous Region (Other); Anhui Provincial Hospital (Other Government); Beijing Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZS-906
Record Dates: First submitted 2016-06-03; First posted 2016-07-25 (Estimated); Last update posted 2022-10-03 (Actual); Status verified 2021-07

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Systemic Lupus Erythematosus; Stable; Relapse Risk; Glucocorticoid Withdrawal
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — Hydroxychloroquine; Glucocorticoids

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Full withdrawal (Experimental): Intervention: 'Drug free'.
  Interventions: Other: Drug free
- GC withdrawal (Experimental): Intervention: 'HCQ' .
  Interventions: Drug: HCQ
- No withdrawal (Experimental): Intervention: 'GC+HCQ' .
  Interventions: Drug: GC+HCQ

INTERVENTIONS:
Other: Drug free — Both Glucocorticoid(GC) and hydroxychloroquine(HCQ) treatment are stopped in stable SLE patients.
  Arms: Full withdrawal
Drug: HCQ — Glucocorticoid(GC) treatment is stopped in stable SLE patients. Hydroxychloroquine (HCQ) is kept as 0.2-0.4g/d
  Other Names: Hydroxychloroquine
  Arms: GC withdrawal
Drug: GC+HCQ — Glucocorticoid(GC) is kept no more than 7.5mg/d. Hydroxychloroquine (HCQ) is kept as 0.2-0.4g/d.
  Other Names: Hydroxychloroquine; Glucocorticoid
  Arms: No withdrawal

SUMMARY:
Whether and when systemic lupus erythematosus (SLE) patients with stable disease should withdraw glucocorticoid (GC)? How about the relapse risk? What are the risk factors for disease flare? All the above are unclear. Long-course GC treatment has a lot of side-effects even in a sustaining low dose. The aim of this study is to explore the relapse risk after GC withdrawal in SLE patients with stable disease more than one year and to establish a predictive model for flare risk stratification.

DETAILED DESCRIPTION:
Systemic lupus erythematosus (SLE) is a chronic autoimmune disease with a relapsing-remitting course. For patients in remission, glucocorticoid (GC) is used to be maintained in a low dose for a long time in fear of disease flare. Long-term GC could bring a lot of side-effects even in a low dose. Whether and when patients with stable disease should withdraw GC? How about the relapse risk? What are the risk factors for disease flare? All the above remain unclear. The aim of this study is to explore the relapse risk after GC withdrawal in SLE patients with stable disease and to establish a predictive model for risk stratification. Meanwhile the investigators aim to testify the effects of hydroxychloroquine in preventing SLE relapse. This study is an open-labeled randomized controlled clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* SLE diagnosis fulfilled the Systemic Lupus International Collaborating Clinic revision of the American College of Rheumatology Classification Criteria for SLE
* Disease stabilized ≥ 1 year
* SELENA-SLEDAI ≤ 3
* Anti-double strand DNA negative by IF measurement and ≤ 200IU/ml by ELISA method
* Complement 3 (C3) ≥ 0.5*lower limit of the normal range, and fluctuation of the C3 is less than 10% within the last year
* 24 hour urine protein ≤ 0.5g
* Prednisone (or equivalent) ≤ 7.5mg/d for more than 6 months
* No use of immunosuppressants including CsA, MMF, CTX, FK506, LEF, MTX in recent 6 months. But hydroxychloroquine (HCQ) is permitted and should be in use
* Never use biologic agents including Rituximab, Belimumab, Epratuzumab and so on
* No severe organ involvement in recent 2 years including lupus encephalosis, diffused alveolar hemorrhage, thrombotic thrombocytopenia purpura, rapid progressive glomerulonephritis, severe thrombocytopenia, severe hemolytic anemia, myocardial involvement, myeleterosis or severe peripheral neuropathy

Exclusion Criteria:

* Active SLE
* In pregnancy or breastfeeding, plan for pregnancy
* Plan or has been on a surgery in recent 6 months
* Current infection
* History of malignancy
* Severe organ dysfunction or other complications
* Unable to follow up
* Inappropriate to be enrolled
* Psoriasis, porphyria, arrhythmia or eye diseases that contradict with HCQ usage

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 333 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Percent of subjects with mild to moderate Lupus flare evaluated by modified SELENA-SLEDAI flare index (SFI) | 33 weeks
  The SFI includes three elements: the SELENA-SLEDAI score (range 0 ~105, with 0 indicating inactive disease and ); an assessment of new or worsening disease activity, medication changes, and hospitalizations that not captured with the use of the SLEDAI; and the score on the physician's global-assessment (PGA) visual-analogue scale (range, 0 to 3, 1=mild, 2=moderate, 3=severe); Mild to moderate flare by SFI is defined as appearance of one of the following: a change in SLEDAI>3 points but≤12 points; or new onset/worse of cutaneous/ mucosal injury (discoid, photosensitivity, profundus, cutaneous vasculitis, bullous lupus, Nasopharyngeal ulcers), serositis (pleuritis and/or pericarditis), arthritis, SLE associated fever; or the need to increase prednisone dosage to no more than 0.5 mg/kg/day; or the need to add hydroxychloroquine or NSAIDs with no increase in the dose GC; or an increment of PGA ranges from 1.0 to 2.5.

SECONDARY OUTCOMES:
Percent of subjects with a SELENA-SLEDAI maintaining at <4 points | 33 weeks
Mean change in PGA | 33 weeks
  The PGA is a visual analog scale scored from 0 to 3. A score of 1 corresponds to mild lupus disease activity; A score of 2 correlates with moderate disease activity and a score of 3 with severe disease activity
• Percent of subjects with at least one B in any system evaluated with The British Isles Lupus Activity Group (BILAG) scoring system | 33 weeks
  BILAG includes 9 systems (constitutional, mucocutaneous, neuropsychiatric, musculoskeletal, cardiorespiratory, gastrointestinal, ophthalmic, renal and haematological). A to E scoring is based on the physician's intention to treat: Grade A: treatment requiring any of the following 1) high dose oral glucocorticoids, eg: prednisolone>20mg/day; 2) intravenous pulse glucocorticoids, eg: pulse methylprednisolone ≥ 500 mg；3)systemic immunomodulators (include biologicals, immunoglobulins and plasmapheresis)；4) therapeutic high dose anticoagulation, eg: warfarin INR 3 - 4; Grade B: treatment requiring any of the following treatment:1) low dose oral glucocorticoids, eg: prednisolone ≤ 20mg/day; 2) intramuscular or intra-articular or soft tissue glucocorticoids injection; 3) topical glucocorticoids;4) topical immunomodulators; 5) antimalarials or thalidomide;6) symptomatic therapy; eg: NSAIDs; Grade C: mild disease; Grade D: inactive now but previously affected; Grade E: systems never involved

CONTACTS AND LOCATIONS:
Overall Officials: Xuan Zhang, MD, Principal Investigator — Peking Union Medical College Hospital; Xuan Zhang, MD, Study Chair — Peking Union Medical College Hospital
Locations (5):
- China (5):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - People's Hospital of Xinjiang Uygur Autonomous Region, Ürümqi, Xinjiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fei Y, Zhao L, Wu L, Zuo X, Li R, Cheng J, Luo H, Wu X, Sun L, Xu J, Zhu Y, Wang Y, Chen Z, Li X, Wang X, Zhang X; PRESS study team. Evaluation and prediction of relapse risk in stable systemic lupus erythematosus patients after glucocorticoid withdrawal (PRESS): an open-label, multicentre, non-inferiority, randomised controlled study in China. Ann Rheum Dis. 2025 Feb;84(2):274-283. doi: 10.1136/ard-2024-225826. Epub 2025 Jan 2. PMID 39919900